CLINICAL TRIAL: NCT01256125
Title: Therapeutic Effects of Allogene MSCs Transplantation in Patients With Chronic Liver Diseases Through Peripheral Vein.
Brief Title: Allogene MSCs Transplantation in Patients With Chronic Liver Diseases Through Peripheral Vein.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Zhi-liang Gao, 3rd Affiliated Hospital of Sun Yat-sen University
Other Study IDs: SunYat-sen U 11-5-1
Record Dates: First submitted 2010-12-07; First posted 2010-12-08 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-10

CONDITIONS: Allogene MSCs Transplantation; Chronic Liver Diseases Patients; Peripheral Vein
Keywords: allogene MSCs; transplantation; chronic liver diseases; peripheral vein

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Allogene MSCs transplantation: Allogene MSCs transplantation were performed in patients with chronic liver diseases through peripheral vein plus the same medical treatments.
- control: only medical treatments were performed in patients with chronic liver diseases.

SUMMARY:
Allogene MSCs transplantation will be performed in patients with chronic liver diseases through peripheral vein and therapeutic effects including short-term effects and long-term follow-up will be compared and investigated.

ELIGIBILITY:
Inclusion Criteria:

1. chronic liver diseases including: viral hepatitis, alcoholic liver disease, autoimmune liver disease.
2. age: 15-65 years old.

Exclusion Criteria:

1. pregnant women and women in lactation.
2. other systems and organs disfunction
3. space-occupying lesion were found in liver.
4. concurrent infection with HIV and other immunodeficiency diseases.
5. DIC and active bleeding were confirmed.

Ages: 15 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic liver diseases including: viral hepatitis, alcoholic liver disease, autoimmune liver disease and so on.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-10

PRIMARY OUTCOMES:
Short-term therapeutic effects at 1-8 weeks after Allogene MSCs transplantation through peripheral vein. | 1-8 weeks after transplantation

SECONDARY OUTCOMES:
Long-term follow-up of Allogene MSCs transplantation through peripheral vein. | 3-60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Infectious Diseases, 3rd Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China